CLINICAL TRIAL: NCT05723796
Title: Study of Nasal Mucosa Histopathological Changes in Patients With Chronic Hypersensitivity Pneumonitis
Brief Title: Study of Nasal Mucosa Histopathological Changes in Chronic Hypersensitivity Pneumonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Kamal Ibrahim Hassan, Assistant Professor of pulmonology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD-138-2021
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hypersensitivity Pneumonitis; Nasal Mucosal Disorder
Keywords: hypersensitivity pneumonitis; nasal mucosa histopaholgical changes
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic HP patients (Experimental)
  Interventions: Procedure: nasal endoscopy

INTERVENTIONS:
Procedure: nasal endoscopy — nasal endoscopy and mucosal biopsy

SUMMARY:
Background:Hypersensitivity pneumonitis (HP) is an interstitial lung disease that develops after inhalation of organic or inorganic antigens in susceptible individuals. The nasal mucosa is constantly exposed to these antigens that can irritate the respiratory mucosa.

Objectives: to assess the burden of sinonasal symptoms in HP patients and to evaluate the nasal histopathology in those patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients with clinical and radiological features of HP

Exclusion Criteria:

* respiratory failure
* patients on anticoagulants

Ages: 29 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
percentage of patients with HP developed nasal mucosa granuloma and lymphocytic infiltrations as detected by nasal endoscopy | 6 months
  nasal endoscopy and nasal mucosa biopsy was done for all patients to measure the % of patients with nasal granuloma and lymphocytic infiltrations

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy school of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akl Y, Ibrahim EK, Algarf TM, Mostafa RR, Abdel-Hamid HM, Muhammed AI. Study of nasal mucosa histopathological changes in patients with hypersensitivity pneumonitis. Sci Rep. 2023 May 31;13(1):8868. doi: 10.1038/s41598-023-35871-5. PMID 37258647